CLINICAL TRIAL: NCT03934203
Title: Thorough QT Study to Evaluate the Effects of BI 409306 as Single Dose on Cardiac Safety Parameters in Healthy Male and Female Subjects. A Randomized, Placebo Controlled, Double-blind, Five-period Crossover Study With (Open-label) Moxifloxacin as Positive Control
Brief Title: This Study in Healthy Men and Women Tests Whether BI 409306 Has an Effect on the ECG (Thorough QT Study)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1289-0038; 2018-001335-44 (EudraCT Number)
Record Dates: First submitted 2019-04-30; First posted 2019-05-01 (Actual); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-08

CONDITIONS: Healthy
MeSH Terms: interventions — BI 409306; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (15):
- H/L/P/P/M treatment sequence (Experimental): In this randomized, placebo-controlled, 5-period crossover trial participants were randomized to one of 15 possible treatment sequences based on a balanced, Prescott triple Latin square design. Treatments administered were 50 mg BI 409306 administered orally as a single dose (1 film-coated tablet plus 4 film-coated placebo tablets), 250 mg BI 409306 administered orally as a single dose (5 film-coated tablets), 400 mg moxifloxacin administered orally as a single dose (1 film-coated tablet), Placebo 1 and Placebo 2 both administered orally as a single dose (5 film-coated tablets). In all treatment periods tablets were taken with 240 milliliter of water after an overnight fast of at least 10 hours on day 1 of the treatment period. The trial was double-blind for placebo and BI 409306, but open-label for moxifloxacin. A washout period of least 6 days was adhered to between drug administrations. L=50 mg BI 409306, H=250 mg BI 409306, M= 400 mg moxifloxacin, P=Placebo 1/Placebo 2.
  Interventions: Drug: BI 409306; Drug: Moxifloxacin; Drug: Placebo matching to BI 409306
- H/M/P/P/L treatment sequence (Experimental): In this randomized, placebo-controlled, 5-period crossover trial participants were randomized to one of 15 possible treatment sequences based on a balanced, Prescott triple Latin square design. Treatments administered were 50 mg BI 409306 administered orally as a single dose (1 film-coated tablet plus 4 film-coated placebo tablets), 250 mg BI 409306 administered orally as a single dose (5 film-coated tablets), 400 mg moxifloxacin administered orally as a single dose (1 film-coated tablet), Placebo 1 and Placebo 2 both administered orally as a single dose (5 film-coated tablets). In all treatment periods tablets were taken with 240 milliliter of water after an overnight fast of at least 10 hours on day 1 of the treatment period. The trial was double-blind for placebo and BI 409306, but open-label for moxifloxacin. A washout period of least 6 days was adhered to between drug administrations. L=50 mg BI 409306, H=250 mg BI 409306, M= 400 mg moxifloxacin, P=Placebo 1/Placebo 2.
  Interventions: Drug: BI 409306; Drug: Moxifloxacin; Drug: Placebo matching to BI 409306
- H/P/P/M/L treatment sequence (Experimental): In this randomized, placebo-controlled, 5-period crossover trial participants were randomized to one of 15 possible treatment sequences based on a balanced, Prescott triple Latin square design. Treatments administered were 50 mg BI 409306 administered orally as a single dose (1 film-coated tablet plus 4 film-coated placebo tablets), 250 mg BI 409306 administered orally as a single dose (5 film-coated tablets), 400 mg moxifloxacin administered orally as a single dose (1 film-coated tablet), Placebo 1 and Placebo 2 both administered orally as a single dose (5 film-coated tablets). In all treatment periods tablets were taken with 240 milliliter of water after an overnight fast of at least 10 hours on day 1 of the treatment period. The trial was double-blind for placebo and BI 409306, but open-label for moxifloxacin. A washout period of least 6 days was adhered to between drug administrations. L=50 mg BI 409306, H=250 mg BI 409306, M= 400 mg moxifloxacin, P=Placebo 1/Placebo 2.
  Interventions: Drug: BI 409306; Drug: Moxifloxacin; Drug: Placebo matching to BI 409306
- L/M/H/P/P treatment sequence (Experimental): In this randomized, placebo-controlled, 5-period crossover trial participants were randomized to one of 15 possible treatment sequences based on a balanced, Prescott triple Latin square design. Treatments administered were 50 mg BI 409306 administered orally as a single dose (1 film-coated tablet plus 4 film-coated placebo tablets), 250 mg BI 409306 administered orally as a single dose (5 film-coated tablets), 400 mg moxifloxacin administered orally as a single dose (1 film-coated tablet), Placebo 1 and Placebo 2 both administered orally as a single dose (5 film-coated tablets). In all treatment periods tablets were taken with 240 milliliter of water after an overnight fast of at least 10 hours on day 1 of the treatment period. The trial was double-blind for placebo and BI 409306, but open-label for moxifloxacin. A washout period of least 6 days was adhered to between drug administrations. L=50 mg BI 409306, H=250 mg BI 409306, M= 400 mg moxifloxacin, P=Placebo 1/Placebo 2.
  Interventions: Drug: BI 409306; Drug: Moxifloxacin; Drug: Placebo matching to BI 409306
- L/P/H/M/P treatment sequence (Experimental): In this randomized, placebo-controlled, 5-period crossover trial participants were randomized to one of 15 possible treatment sequences based on a balanced, Prescott triple Latin square design. Treatments administered were 50 mg BI 409306 administered orally as a single dose (1 film-coated tablet plus 4 film-coated placebo tablets), 250 mg BI 409306 administered orally as a single dose (5 film-coated tablets), 400 mg moxifloxacin administered orally as a single dose (1 film-coated tablet), Placebo 1 and Placebo 2 both administered orally as a single dose (5 film-coated tablets). In all treatment periods tablets were taken with 240 milliliter of water after an overnight fast of at least 10 hours on day 1 of the treatment period. The trial was double-blind for placebo and BI 409306, but open-label for moxifloxacin. A washout period of least 6 days was adhered to between drug administrations. L=50 mg BI 409306, H=250 mg BI 409306, M= 400 mg moxifloxacin, P=Placebo 1/Placebo 2.
  Interventions: Drug: BI 409306; Drug: Moxifloxacin; Drug: Placebo matching to BI 409306
- L/P/M/H/P treatment sequence (Experimental): In this randomized, placebo-controlled, 5-period crossover trial participants were randomized to one of 15 possible treatment sequences based on a balanced, Prescott triple Latin square design. Treatments administered were 50 mg BI 409306 administered orally as a single dose (1 film-coated tablet plus 4 film-coated placebo tablets), 250 mg BI 409306 administered orally as a single dose (5 film-coated tablets), 400 mg moxifloxacin administered orally as a single dose (1 film-coated tablet), Placebo 1 and Placebo 2 both administered orally as a single dose (5 film-coated tablets). In all treatment periods tablets were taken with 240 milliliter of water after an overnight fast of at least 10 hours on day 1 of the treatment period. The trial was double-blind for placebo and BI 409306, but open-label for moxifloxacin. A washout period of least 6 days was adhered to between drug administrations. L=50 mg BI 409306, H=250 mg BI 409306, M= 400 mg moxifloxacin, P=Placebo 1/Placebo 2.
  Interventions: Drug: BI 409306; Drug: Moxifloxacin; Drug: Placebo matching to BI 409306
- M/H/P/L/P treatment sequence (Experimental): In this randomized, placebo-controlled, 5-period crossover trial participants were randomized to one of 15 possible treatment sequences based on a balanced, Prescott triple Latin square design. Treatments administered were 50 mg BI 409306 administered orally as a single dose (1 film-coated tablet plus 4 film-coated placebo tablets), 250 mg BI 409306 administered orally as a single dose (5 film-coated tablets), 400 mg moxifloxacin administered orally as a single dose (1 film-coated tablet), Placebo 1 and Placebo 2 both administered orally as a single dose (5 film-coated tablets). In all treatment periods tablets were taken with 240 milliliter of water after an overnight fast of at least 10 hours on day 1 of the treatment period. The trial was double-blind for placebo and BI 409306, but open-label for moxifloxacin. A washout period of least 6 days was adhered to between drug administrations. L=50 mg BI 409306, H=250 mg BI 409306, M= 400 mg moxifloxacin, P=Placebo 1/Placebo 2.
  Interventions: Drug: BI 409306; Drug: Moxifloxacin; Drug: Placebo matching to BI 409306
- M/L/P/H/P treatment sequence (Experimental): In this randomized, placebo-controlled, 5-period crossover trial participants were randomized to one of 15 possible treatment sequences based on a balanced, Prescott triple Latin square design. Treatments administered were 50 mg BI 409306 administered orally as a single dose (1 film-coated tablet plus 4 film-coated placebo tablets), 250 mg BI 409306 administered orally as a single dose (5 film-coated tablets), 400 mg moxifloxacin administered orally as a single dose (1 film-coated tablet), Placebo 1 and Placebo 2 both administered orally as a single dose (5 film-coated tablets). In all treatment periods tablets were taken with 240 milliliter of water after an overnight fast of at least 10 hours on day 1 of the treatment period. The trial was double-blind for placebo and BI 409306, but open-label for moxifloxacin. A washout period of least 6 days was adhered to between drug administrations. L=50 mg BI 409306, H=250 mg BI 409306, M= 400 mg moxifloxacin, P=Placebo 1/Placebo 2.
  Interventions: Drug: BI 409306; Drug: Moxifloxacin; Drug: Placebo matching to BI 409306
- M/P/H/P/L treatment sequence (Experimental): In this randomized, placebo-controlled, 5-period crossover trial participants were randomized to one of 15 possible treatment sequences based on a balanced, Prescott triple Latin square design. Treatments administered were 50 mg BI 409306 administered orally as a single dose (1 film-coated tablet plus 4 film-coated placebo tablets), 250 mg BI 409306 administered orally as a single dose (5 film-coated tablets), 400 mg moxifloxacin administered orally as a single dose (1 film-coated tablet), Placebo 1 and Placebo 2 both administered orally as a single dose (5 film-coated tablets). In all treatment periods tablets were taken with 240 milliliter of water after an overnight fast of at least 10 hours on day 1 of the treatment period. The trial was double-blind for placebo and BI 409306, but open-label for moxifloxacin. A washout period of least 6 days was adhered to between drug administrations. L=50 mg BI 409306, H=250 mg BI 409306, M= 400 mg moxifloxacin, P=Placebo 1/Placebo 2.
  Interventions: Drug: BI 409306; Drug: Moxifloxacin; Drug: Placebo matching to BI 409306
- P/H/L/M/P treatment sequence (Experimental): In this randomized, placebo-controlled, 5-period crossover trial participants were randomized to one of 15 possible treatment sequences based on a balanced, Prescott triple Latin square design. Treatments administered were 50 mg BI 409306 administered orally as a single dose (1 film-coated tablet plus 4 film-coated placebo tablets), 250 mg BI 409306 administered orally as a single dose (5 film-coated tablets), 400 mg moxifloxacin administered orally as a single dose (1 film-coated tablet), Placebo 1 and Placebo 2 both administered orally as a single dose (5 film-coated tablets). In all treatment periods tablets were taken with 240 milliliter of water after an overnight fast of at least 10 hours on day 1 of the treatment period. The trial was double-blind for placebo and BI 409306, but open-label for moxifloxacin. A washout period of least 6 days was adhered to between drug administrations. L=50 mg BI 409306, H=250 mg BI 409306, M= 400 mg moxifloxacin, P=Placebo 1/Placebo 2.
  Interventions: Drug: BI 409306; Drug: Moxifloxacin; Drug: Placebo matching to BI 409306
- P/H/L/P/M treatment sequence (Experimental): In this randomized, placebo-controlled, 5-period crossover trial participants were randomized to one of 15 possible treatment sequences based on a balanced, Prescott triple Latin square design. Treatments administered were 50 mg BI 409306 administered orally as a single dose (1 film-coated tablet plus 4 film-coated placebo tablets), 250 mg BI 409306 administered orally as a single dose (5 film-coated tablets), 400 mg moxifloxacin administered orally as a single dose (1 film-coated tablet), Placebo 1 and Placebo 2 both administered orally as a single dose (5 film-coated tablets). In all treatment periods tablets were taken with 240 milliliter of water after an overnight fast of at least 10 hours on day 1 of the treatment period. The trial was double-blind for placebo and BI 409306, but open-label for moxifloxacin. A washout period of least 6 days was adhered to between drug administrations. L=50 mg BI 409306, H=250 mg BI 409306, M= 400 mg moxifloxacin, P=Placebo 1/Placebo 2.
  Interventions: Drug: BI 409306; Drug: Moxifloxacin; Drug: Placebo matching to BI 409306
- P/L/M/P/H treatment sequence (Experimental): In this randomized, placebo-controlled, 5-period crossover trial participants were randomized to one of 15 possible treatment sequences based on a balanced, Prescott triple Latin square design. Treatments administered were 50 mg BI 409306 administered orally as a single dose (1 film-coated tablet plus 4 film-coated placebo tablets), 250 mg BI 409306 administered orally as a single dose (5 film-coated tablets), 400 mg moxifloxacin administered orally as a single dose (1 film-coated tablet), Placebo 1 and Placebo 2 both administered orally as a single dose (5 film-coated tablets). In all treatment periods tablets were taken with 240 milliliter of water after an overnight fast of at least 10 hours on day 1 of the treatment period. The trial was double-blind for placebo and BI 409306, but open-label for moxifloxacin. A washout period of least 6 days was adhered to between drug administrations. L=50 mg BI 409306, H=250 mg BI 409306, M= 400 mg moxifloxacin, P=Placebo 1/Placebo 2.
  Interventions: Drug: BI 409306; Drug: Moxifloxacin; Drug: Placebo matching to BI 409306
- P/M/P/L/H treatment sequence (Experimental): In this randomized, placebo-controlled, 5-period crossover trial participants were randomized to one of 15 possible treatment sequences based on a balanced, Prescott triple Latin square design. Treatments administered were 50 mg BI 409306 administered orally as a single dose (1 film-coated tablet plus 4 film-coated placebo tablets), 250 mg BI 409306 administered orally as a single dose (5 film-coated tablets), 400 mg moxifloxacin administered orally as a single dose (1 film-coated tablet), Placebo 1 and Placebo 2 both administered orally as a single dose (5 film-coated tablets). In all treatment periods tablets were taken with 240 milliliter of water after an overnight fast of at least 10 hours on day 1 of the treatment period. The trial was double-blind for placebo and BI 409306, but open-label for moxifloxacin. A washout period of least 6 days was adhered to between drug administrations. L=50 mg BI 409306, H=250 mg BI 409306, M= 400 mg moxifloxacin, P=Placebo 1/Placebo 2.
  Interventions: Drug: BI 409306; Drug: Moxifloxacin; Drug: Placebo matching to BI 409306
- P/P/L/H/M treatment sequence (Experimental): In this randomized, placebo-controlled, 5-period crossover trial participants were randomized to one of 15 possible treatment sequences based on a balanced, Prescott triple Latin square design. Treatments administered were 50 mg BI 409306 administered orally as a single dose (1 film-coated tablet plus 4 film-coated placebo tablets), 250 mg BI 409306 administered orally as a single dose (5 film-coated tablets), 400 mg moxifloxacin administered orally as a single dose (1 film-coated tablet), Placebo 1 and Placebo 2 both administered orally as a single dose (5 film-coated tablets). In all treatment periods tablets were taken with 240 milliliter of water after an overnight fast of at least 10 hours on day 1 of the treatment period. The trial was double-blind for placebo and BI 409306, but open-label for moxifloxacin. A washout period of least 6 days was adhered to between drug administrations. L=50 mg BI 409306, H=250 mg BI 409306, M= 400 mg moxifloxacin, P=Placebo 1/Placebo 2.
  Interventions: Drug: BI 409306; Drug: Moxifloxacin; Drug: Placebo matching to BI 409306
- P/P/M/L/H treatment sequence (Experimental): In this randomized, placebo-controlled, 5-period crossover trial participants were randomized to one of 15 possible treatment sequences based on a balanced, Prescott triple Latin square design. Treatments administered were 50 mg BI 409306 administered orally as a single dose (1 film-coated tablet plus 4 film-coated placebo tablets), 250 mg BI 409306 administered orally as a single dose (5 film-coated tablets), 400 mg moxifloxacin administered orally as a single dose (1 film-coated tablet), Placebo 1 and Placebo 2 both administered orally as a single dose (5 film-coated tablets). In all treatment periods tablets were taken with 240 milliliter of water after an overnight fast of at least 10 hours on day 1 of the treatment period. The trial was double-blind for placebo and BI 409306, but open-label for moxifloxacin. A washout period of least 6 days was adhered to between drug administrations. L=50 mg BI 409306, H=250 mg BI 409306, M= 400 mg moxifloxacin, P=Placebo 1/Placebo 2.
  Interventions: Drug: BI 409306; Drug: Moxifloxacin; Drug: Placebo matching to BI 409306

INTERVENTIONS:
Drug: BI 409306 — Film-coated tablet
Drug: Moxifloxacin — Film-coated tablet
  Other Names: Avalox®
Drug: Placebo matching to BI 409306 — Film-coated tablet

SUMMARY:
The primary objective of this trial is to assess the effect of BI 409306 on the QT/QTc interval in healthy male and female volunteers as measured by the QTcF change from baseline compared with placebo.

Secondary objectives are to show the assay sensitivity of the trial, by reproducing the typical effect of the positive control moxifloxacin on the QT/QTc interval, and to assess the effect of BI 409306 on heart rate.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects according to the assessment of the investigator, based on a complete medical history including a physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead single Electrocardiogram (ECG) and 12-lead Holter Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 50 years (incl.)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with Good clinical practice (GCP) and local legislation
* Male subjects, or female subjects who meet any of the following criteria starting from at least 30 days before the first administration of trial medication and until 30 days after trial completion:

  * Use of adequate contraception, e.g. non-hormonal intrauterine device plus condom
  * Sexually abstinent
  * A vasectomised sexual partner (vasectomy at least 1 year prior to enrolment)
  * Surgically sterilised (including hysterectomy)
  * Postmenopausal, defined as at least 1 year of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous levels of FSH above 40 U/L and estradiol below 30 ng/L is confirmatory)

Exclusion Criteria:

* Any finding in the medical examination (including Blood Pressure (BP), Pulse Rate (PR) or Electrocardiogram (ECG)) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 100 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Further exclusion criteria apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2019-09-06 (Actual); Study Completion 2019-09-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization). For more details refer to: http://trials.boehringer-ingelheim.com/

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, placebo-controlled, double-blind trial with crossover design with 5 treatment periods, 15 treatment sequences based on a balanced, Prescott triple Latin square design with a wash-out period of at least 6 days between treatments: 50 mg BI 409306, 250 mg BI 409306, 400 mg moxifloxacin (positive control, open-label), placebo (2 periods).
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated. Abbreviation: mg=milligram.
  There was a washout period of at least 6 days between treatments.
Period: Overall Study
Arm/Group | H/L/P/P/M Treatment Sequence | H/M/P/P/L Treatment Sequence | H/P/P/M/L Treatment Sequence | L/M/H/P/P Treatment Sequence | L/P/H/M/P Treatment Sequence | L/P/M/H/P Treatment Sequence | M/H/P/L/P Treatment Sequence | M/L/P/H/P Treatment Sequence | M/P/H/P/L Treatment Sequence | P/H/L/M/P Treatment Sequence | P/H/L/P/M Treatment Sequence | P/L/M/P/H Treatment Sequence | P/M/P/L/H Treatment Sequence | P/P/L/H/M Treatment Sequence | P/P/M/L/H Treatment Sequence
Started | 3 | 3 | 3 | 3 | 4 | 3 | 4 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 2 | 3 | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 3
Not Completed | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): This participant set included all randomized participants who received at least one dose of any trial medication.
Groups:
- Overall Study: Total number of participants randomized and treated in this randomized, placebo-controlled, 5-period crossover trial where participants were randomized to one of 15 possible treatment sequences based on a balanced, Prescott triple Latin square design. Treatments administered were 50 milligram (mg) BI 409306 administered orally as a single dose (1 film-coated tablet plus 4 film-coated placebo tablets), 250 mg BI 409306 administered orally as a single dose (5 film-coated tablets), 400 mg moxifloxacin administered orally as a single dose (1 film-coated tablet), Placebo 1 and Placebo 2 both administered orally as a single dose (5 film-coated tablets). In all treatment periods tablets were taken with 240 milliliter of water after an overnight fast of at least 10 hours on day 1 of the treatment period. The trial was double-blind for placebo and BI 409306, but open-label for moxifloxacin. A washout period of least 6 days was adhered to between drug administrations.
Arm/Group | Overall Study
Number analyzed (Participants) | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 47
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 46
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in QTcF at That Timepoint Between 20 Minutes to 24 Hours After Drug Administration Where the Difference of Means in QTcF Changes From Baseline Between 50 Milligram (mg) BI 409306 and Placebo Takes Its Maximum
Description: QTcF is the QT interval (Electrocardiogram (ECG) interval from the beginning of the QRS complex to the end of the T wave) corrected using Fridericia's formula. Change from baseline in QTcF at that timepoint between 20 minutes to 24 hours after drug administration where the difference of means in QTcF changes from baseline between 50 mg BI 409306 and placebo takes its maximum.
  A linear mixed-effects model for repeated measurements based on Schall and Ring (MMRM) was fitted to the observations for 50 mg BI 409306 and the 2 placebo periods.
  Total number of participants per treatment and timepoint can be lower than 47 due to participants having left their treatment sequence before being exposed to the respective treatment, or due to exclusion of individual participant ECG data at timepoints affected by ECG-relevant important protocol deviations.
Time Frame: Baseline, 20 minutes (min), 40 min, 1 hour (h), 1 h 30 min, 2 h, 2 h 30 min, 3 h, 4 h, 8 h, 12 h, 24 h after study drug administration
Population: ECG Set: This participant set included all randomized participants who received at least one dose of any trial medication and who had at least one on-treatment value for at least one electrocardiogram (ECG) endpoint, which was not excluded due to ECG-relevant important protocol deviations (e.g. the use of pro-arrhythmic medications).
Measure: Least Squares Mean (Standard Error); unit: milliseconds
Units Other Than Participants: Observations
Groups:
- Placebo to BI 409306 in 2 Periods: Placebo administered orally as a single dose (5 film-coated tablets) taken with 240 milliliter of water after an overnight fast of at least 10 hours on day 1 of the treatment period. Placebo was administered in two treatment periods.
- 50 Milligram (mg) BI 409306: 50 milligram (mg) BI 409306 administered orally as a single dose (1 film-coated tablet plus 4 film-coated placebo tablets) taken with 240 milliliter of water after an overnight fast of at least 10 hours on day 1 of the treatment period.
Arm/Group | Placebo to BI 409306 in 2 Periods | 50 Milligram (mg) BI 409306
Number analyzed (Participants) | 47 | 45
Number analyzed (Observations) | 1000 | 493
milliseconds
  20 min after drug intake=timepoint of maximum: number analyzed (Observations) | 90 | 45
  20 min after drug intake=timepoint of maximum | -1.5 (0.4) | -0.2 (0.6)
  40 minutes after drug intake: number analyzed (Observations) | 91 | 45
  40 minutes after drug intake | -1.0 (0.4) | -0.8 (0.6)
  1 hour after drug intake: number analyzed (Observations) | 91 | 45
  1 hour after drug intake | -0.5 (0.4) | 0.3 (0.6)
  1 hour and 30 minutes after drug intake: number analyzed (Participants) | 47 | 43
  1 hour and 30 minutes after drug intake: number analyzed (Observations) | 91 | 43
  1 hour and 30 minutes after drug intake | -0.1 (0.5) | -0.4 (0.7)
  2 hours after drug intake: number analyzed (Observations) | 91 | 45
  2 hours after drug intake | -0.1 (0.5) | -0.3 (0.7)
  2 hours and 30 minutes after drug intake: number analyzed (Observations) | 91 | 45
  2 hours and 30 minutes after drug intake | -2.0 (0.5) | -1.7 (0.7)
  3 hours after drug intake: number analyzed (Observations) | 91 | 45
  3 hours after drug intake | 0.4 (0.5) | -0.2 (0.7)
  4 hours after drug intake: number analyzed (Observations) | 91 | 45
  4 hours after drug intake | 1.0 (0.6) | 0.0 (0.8)
  8 hours after drug intake: number analyzed (Observations) | 91 | 45
  8 hours after drug intake | -7.0 (0.7) | -7.3 (0.9)
  12 hours after drug intake: number analyzed (Observations) | 91 | 45
  12 hours after drug intake | -1.0 (0.7) | -1.0 (1.0)
  24 hours after drug intake: number analyzed (Observations) | 91 | 45
  24 hours after drug intake | -6.4 (0.6) | -5.8 (0.8)
Statistical Analysis 1: Comparison: Placebo to BI 409306 in 2 Periods vs 50 Milligram (mg) BI 409306; MMRM was fitted to observations for 50 mg BI 409306 and the 2 placebo periods. MMRM with covariates 'period baseline', 'participant baseline' (=arithmetic mean of respective period baselines), fixed categorical effects 'treatment', 'period', and 'time', interaction terms 'period baseline-by-time', 'participant baseline-by-time', 'treatment-by-time', and 'period-by-time', 'participant' (random effect), and time within period as repeated measures per participant (covariance matrix=Unstructured); Test type: Other — The null hypothesis was 'The mean difference in the QTcF changes from baseline between 50 mg BI 409306 and placebo is greater than or equal to 10 milliseconds at least for one timepoint after dosing.' The one-sided tests were performed at the 5% level; due to the symmetry of the normal distribution 2-sided 90% confidence intervals for the differences of adjusted means per timepoint were used; Mixed Models Analysis; Restricted maximum likelihood estimation and Kenward-Roger method to adjust standard errors and estimate denominator degrees of freedom; Difference of adjusted means = 1.3, 90% CI 2-sided [0.2 to 2.4], Standard Error of Mean 0.7 — Maximum difference of adjusted means was calculated as BI 409306 - placebo at 20 minutes after drug intake

2. Primary Outcome: Change From Baseline in QTcF at That Timepoint Between 20 Minutes to 24 Hours After Drug Administration Where the Difference of Means in QTcF Changes From Baseline Between 250 Milligram (mg) BI 409306 and Placebo Takes Its Maximum
Description: QTcF is the QT interval (Electrocardiogram (ECG) interval from the beginning of the QRS complex to the end of the T wave) corrected using Fridericia's formula. Change from baseline in QTcF at that timepoint between 20 minutes to 24 hours after drug administration where the difference of means in QTcF changes from baseline between 250 mg BI 409306 and placebo takes its maximum.
  A linear mixed-effects model for repeated measurements based on Schall and Ring (MMRM) was fitted to the observations for 250 mg BI 409306 and the 2 placebo periods.
  Total number of participants per treatment and timepoint can be lower than 47 due to participants having left their treatment sequence before being exposed to the respective treatment, or due to exclusion of individual participant ECG data at timepoints affected by ECG-relevant important protocol deviations.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: milliseconds
Units Other Than Participants: Observations
Groups:
- 250 Milligram (mg) BI 409306: 250 mg BI 409306 administered orally as a single dose (5 film-coated tablets) taken with 240 milliliter of water after an overnight fast of at least 10 hours on day 1 of the treatment period.
Arm/Group | Placebo to BI 409306 in 2 Periods | 250 Milligram (mg) BI 409306
Number analyzed (Participants) | 47 | 46
Number analyzed (Observations) | 1000 | 505
milliseconds
  20 minutes after drug intake: number analyzed (Participants) | 47 | 45
  20 minutes after drug intake: number analyzed (Observations) | 90 | 45
  20 minutes after drug intake | -1.4 (0.5) | 2.5 (0.6)
  40 minutes after drug intake= timepoint of maximum: number analyzed (Observations) | 91 | 46
  40 minutes after drug intake= timepoint of maximum | -1.0 (0.5) | 4.7 (0.7)
  1 hour after drug intake: number analyzed (Observations) | 91 | 46
  1 hour after drug intake | -0.4 (0.5) | 3.3 (0.7)
  1 hour and 30 minutes after drug intake: number analyzed (Observations) | 91 | 46
  1 hour and 30 minutes after drug intake | -0.0 (0.5) | 2.7 (0.7)
  2 hours after drug intake: number analyzed (Observations) | 91 | 46
  2 hours after drug intake | -0.1 (0.5) | 1.7 (0.7)
  2 hours and 30 minutes after drug intake: number analyzed (Observations) | 91 | 46
  2 hours and 30 minutes after drug intake | -1.9 (0.6) | -0.7 (0.8)
  3 hours after drug intake: number analyzed (Observations) | 91 | 46
  3 hours after drug intake | 0.4 (0.5) | 1.3 (0.7)
  4 hours after drug intake: number analyzed (Observations) | 91 | 46
  4 hours after drug intake | 1.0 (0.5) | 1.6 (0.8)
  8 hours after drug intake: number analyzed (Observations) | 91 | 46
  8 hours after drug intake | -6.8 (0.7) | -7.3 (0.9)
  12 hours after drug intake: number analyzed (Observations) | 91 | 46
  12 hours after drug intake | -0.9 (0.7) | -0.9 (1.0)
  24 hours after drug intake: number analyzed (Observations) | 91 | 46
  24 hours after drug intake | -6.3 (0.6) | -5.7 (0.8)
Statistical Analysis 1: Comparison: Placebo to BI 409306 in 2 Periods vs 250 Milligram (mg) BI 409306; MMRM was fitted to observations for 250 mg BI 409306 and the 2 placebo periods. MMRM with covariates 'period baseline', 'participant baseline' (=arithmetic mean of respective period baselines), fixed categorical effects 'treatment', 'period', and 'time', interaction terms 'period baseline-by-time', 'participant baseline-by-time', 'treatment-by-time', and 'period-by-time', 'participant' (random effect), and time within period as repeated measures per participant (covariance matrix=Unstructured); Test type: Other — The null hypothesis was 'The mean difference in the QTcF changes from baseline between 250 mg BI 409306 and placebo is greater than or equal to 10 milliseconds at least for one timepoint after dosing.' The one-sided tests were performed at the 5% level; due to the symmetry of the normal distribution 2-sided 90% confidence intervals for the differences of adjusted means per timepoint were used; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Difference of adjusted means = 5.7, 90% CI 2-sided [4.4 to 7.1], Standard Error of Mean 0.8 — Maximum difference of adjusted means was calculated as BI 409306 - placebo at 40 minutes after drug intake

3. Secondary Outcome: Change From Baseline in QTcF at That Timepoint Between 20 Minutes to 24 Hours After Drug Administration Where the Difference of Means in QTcF Changes From Baseline Between Moxifloxacin and Placebo Takes Its Maximum
Description: QTcF is the QT interval (Electrocardiogram (ECG) interval from the beginning of the QRS complex to the end of the T wave) corrected using Fridericia's formula. Change from baseline in QTcF at that timepoint between 20 minutes to 24 hours after drug administration where the difference of means in QTcF changes from baseline between moxifloxacin and placebo takes its maximum.
  A linear mixed-effects model for repeated measurements based on Schall and Ring (MMRM) was fitted to the observations for moxifloxacin and the 2 placebo periods.
  Total number of participants per treatment and timepoint can be lower than 47 due to participants having left their treatment sequence before being exposed to the respective treatment, or due to exclusion of individual participant ECG data at timepoints affected by ECG-relevant important protocol deviations.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: milliseconds
Units Other Than Participants: Observations
Groups:
- 400 Milligram (mg) Moxifloxacin: 400 mg moxifloxacin administered orally as a single dose (1 film-coated tablet) taken with 240 milliliter of water after an overnight fast of at least 10 hours on day 1 of the treatment period.
Arm/Group | Placebo to BI 409306 in 2 Periods | 400 Milligram (mg) Moxifloxacin
Number analyzed (Participants) | 47 | 45
Number analyzed (Observations) | 1000 | 495
milliseconds
  20 min after drug intake: number analyzed (Observations) | 90 | 45
  20 min after drug intake | -1.5 (0.4) | -1.2 (0.6)
  40 minutes after drug intake: number analyzed (Observations) | 91 | 45
  40 minutes after drug intake | -1.0 (0.5) | 7.7 (0.7)
  1 hour after drug intake: number analyzed (Observations) | 91 | 45
  1 hour after drug intake | -0.5 (0.5) | 11.4 (0.7)
  1 h 30 min after drug intake=timepoint of maximum: number analyzed (Observations) | 91 | 45
  1 h 30 min after drug intake=timepoint of maximum | -0.1 (0.5) | 12.0 (0.8)
  2 hours after drug intake: number analyzed (Observations) | 91 | 45
  2 hours after drug intake | -0.1 (0.5) | 11.8 (0.7)
  2 hours and 30 minutes after drug intake: number analyzed (Observations) | 91 | 45
  2 hours and 30 minutes after drug intake | -2.0 (0.6) | 8.4 (0.9)
  3 hours after drug intake: number analyzed (Observations) | 91 | 45
  3 hours after drug intake | 0.4 (0.6) | 11.4 (0.9)
  4 hours after drug intake: number analyzed (Observations) | 91 | 45
  4 hours after drug intake | 1.0 (0.6) | 11.7 (0.9)
  8 hours after drug intake: number analyzed (Observations) | 91 | 45
  8 hours after drug intake | -7.0 (0.7) | 2.3 (1.0)
  12 hours after drug intake: number analyzed (Observations) | 91 | 45
  12 hours after drug intake | -0.9 (0.7) | 5.0 (1.0)
  24 hours after drug intake: number analyzed (Observations) | 91 | 45
  24 hours after drug intake | -6.5 (0.6) | -0.7 (0.9)
Statistical Analysis 1: Comparison: Placebo to BI 409306 in 2 Periods vs 400 Milligram (mg) Moxifloxacin; MMRM was fitted to the observations for moxifloxacin and the 2 placebo periods. MMRM with covariates 'period baseline', 'participant baseline' (=arithmetic mean of respective period baselines), fixed categorical effects 'treatment', 'period', and 'time', interaction terms 'period baseline-by-time', 'participant baseline-by-time', 'treatment-by-time', and 'period-by-time', 'participant' (random effect), and time within period as repeated measures per participant (covariance matrix=Unstructured); Test type: Other — No formal hypotheses were tested; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Difference of adjusted means = 12.1, 90% CI 2-sided [10.5 to 13.6], Standard Error of Mean 0.9 — Maximum difference of adjusted means was calculated as moxifloxacin - placebo at 1 hour and 30 minutes after drug intake

4. Secondary Outcome: Change From Baseline in QTcF at 2 Hours After Drug Administration (Assessment of Assay Sensitivity)
Description: QTcF is the QT interval (Electrocardiogram (ECG) interval from the beginning of the QRS complex to the end of the T wave) corrected using Fridericia's formula. Change from baseline in QTcF at 2 hours after drug administration.
  A linear mixed-effects model for repeated measurements based on Schall and Ring (MMRM) was fitted to the observations for moxifloxacin and the 2 placebo periods.
  Total number of participants per treatment and timepoint can be lower than 47 due to participants having left their treatment sequence before being exposed to the respective treatment, or due to exclusion of individual participant ECG data at timepoints affected by ECG-relevant important protocol deviations.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: milliseconds
Units Other Than Participants: Observations
Arm/Group | Placebo to BI 409306 in 2 Periods | 400 Milligram (mg) Moxifloxacin
Number analyzed (Participants) | 47 | 45
Number analyzed (Observations) | 91 | 45
milliseconds | -0.1 (0.5) | 11.8 (0.7)
Statistical Analysis 1: Comparison: Placebo to BI 409306 in 2 Periods vs 400 Milligram (mg) Moxifloxacin; [analysis description as in outcome 3, analysis 1]; Test type: Other — T-Test based on the results of the MMRM (fitted to the data for all timepoints). The null hypothesis was 'The mean difference in the QTcF changes from baseline between moxifloxacin and placebo is less than or equal to 5 milliseconds at 2 hours after drug administration.'; p = 0.00000000, Mixed Models Analysis — The corresponding alpha-level according to Hochberg's adjustment for mulitplicity was 0.0167; [statistical method as in outcome 1, analysis 1]; Difference of adjusted means = 11.9, 90% CI 2-sided [10.4 to 13.4], Standard Error of Mean 0.9 — Difference of adjusted means was calculated as moxifloxacin - placebo

5. Secondary Outcome: Change From Baseline in QTcF at 3 Hours After Drug Administration (Assessment of Assay Sensitivity)
Description: QTcF is the QT interval (Electrocardiogram (ECG) interval from the beginning of the QRS complex to the end of the T wave) corrected using Fridericia's formula. Change from baseline in QTcF at 3 hours after drug administration.
  A linear mixed-effects model for repeated measurements based on Schall and Ring (MMRM) was fitted to the observations for moxifloxacin and the 2 placebo periods.
  Total number of participants per treatment and timepoint can be lower than 47 due to participants having left their treatment sequence before being exposed to the respective treatment, or due to exclusion of individual participant ECG data at timepoints affected by ECG-relevant important protocol deviations.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: milliseconds
Units Other Than Participants: Observations
Arm/Group | Placebo to BI 409306 in 2 Periods | 400 Milligram (mg) Moxifloxacin
Number analyzed (Participants) | 47 | 45
Number analyzed (Observations) | 91 | 45
milliseconds | 0.4 (0.6) | 11.4 (0.9)
Statistical Analysis 1: Comparison: Placebo to BI 409306 in 2 Periods vs 400 Milligram (mg) Moxifloxacin; [analysis description as in outcome 3, analysis 1]; Test type: Other — T-Test based on the results of the MMRM (fitted to the data for all timepoints). The null hypothesis was 'The mean difference in the QTcF changes from baseline between moxifloxacin and placebo is less than or equal to 5 milliseconds at 3 hours after drug administration.'; p = 0.00000003, Mixed Models Analysis — The corresponding alpha-level according to Hochberg's adjustment for mulitplicity was 0.0250; [statistical method as in outcome 1, analysis 1]; Difference of adjusted means = 11.1, 90% CI 2-sided [9.3 to 12.8], Standard Error of Mean 1.0 — Difference of adjusted means was calculated as moxifloxacin - placebo

6. Secondary Outcome: Change From Baseline in QTcF at 4 Hours After Drug Administration (Assessment of Assay Sensitivity)
Description: QTcF is the QT interval (Electrocardiogram (ECG) interval from the beginning of the QRS complex to the end of the T wave) corrected using Fridericia's formula. Change from baseline in QTcF at 4 hours after drug administration.
  A linear mixed-effects model for repeated measurements based on Schall and Ring (MMRM) was fitted to the observations for moxifloxacin and the 2 placebo periods.
  Total number of participants per treatment and timepoint can be lower than 47 due to participants having left their treatment sequence before being exposed to the respective treatment, or due to exclusion of individual participant ECG data at timepoints affected by ECG-relevant important protocol deviations.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: milliseconds
Units Other Than Participants: Observations
Arm/Group | Placebo to BI 409306 in 2 Periods | 400 Milligram (mg) Moxifloxacin
Number analyzed (Participants) | 47 | 45
Number analyzed (Observations) | 91 | 45
milliseconds | 1.0 (0.6) | 11.7 (0.9)
Statistical Analysis 1: Comparison: Placebo to BI 409306 in 2 Periods vs 400 Milligram (mg) Moxifloxacin; [analysis description as in outcome 3, analysis 1]; Test type: Other — T-Test based on the results of the MMRM (fitted to the data for all timepoints). The null hypothesis was 'The mean difference in the QTcF changes from baseline between moxifloxacin and placebo is less than or equal to 5 milliseconds at 4 hours after drug administration.'; p = 0.00000020, Mixed Models Analysis — The corresponding alpha-level according to Hochberg's adjustment for mulitplicity was 0.050; [statistical method as in outcome 1, analysis 1]; Difference of adjusted means = 10.7, 90% CI 2-sided [8.9 to 12.4], Standard Error of Mean 1.1 — Difference of adjusted means was calculated as moxifloxacin - placebo

7. Secondary Outcome: Change From Baseline in Heart Rate (HR) at That Timepoint Between 20 Minutes to 24 Hours After Drug Administration Where the Difference of Means in Heart Rate Changes From Baseline Between 50 Milligram (mg) BI 409306 and Placebo Takes Its Maximum
Description: Change from baseline in heart rate (HR) at each timepoint between 20 minutes to 24 hours after drug administration where the difference of means in heart rate changes from baseline between 50 milligram (mg) BI 409306 and placebo takes its maximum.
  A linear mixed-effects model for repeated measurements based on Schall and Ring (MMRM) was fitted to the observations for 50 mg BI 409306 and the 2 placebo periods.
  Total number of participants per treatment and timepoint can be lower than 47 due to participants having left their treatment sequence before being exposed to the respective treatment, or due to exclusion of individual participant ECG data at timepoints affected by ECG-relevant important protocol deviations.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: beats / minute
Units Other Than Participants: Observations
Arm/Group | Placebo to BI 409306 in 2 Periods | 50 Milligram (mg) BI 409306
Number analyzed (Participants) | 47 | 45
Number analyzed (Observations) | 1000 | 493
beats / minute
  20 min after drug intake = timepoint of maximum: number analyzed (Observations) | 90 | 45
  20 min after drug intake = timepoint of maximum | 0.6 (0.4) | 3.0 (0.5)
  40 minutes (min) after drug intake: number analyzed (Observations) | 91 | 45
  40 minutes (min) after drug intake | 0.4 (0.4) | 2.5 (0.5)
  1 hour after drug intake: number analyzed (Observations) | 91 | 45
  1 hour after drug intake | 0.5 (0.4) | 1.9 (0.5)
  1 hour and 30 minutes after drug intake: number analyzed (Participants) | 47 | 43
  1 hour and 30 minutes after drug intake: number analyzed (Observations) | 91 | 43
  1 hour and 30 minutes after drug intake | 0.7 (0.4) | 0.8 (0.5)
  2 hours after drug intake: number analyzed (Observations) | 91 | 45
  2 hours after drug intake | 0.9 (0.4) | 0.8 (0.5)
  2 hours and 30 minutes after drug intake: number analyzed (Observations) | 91 | 45
  2 hours and 30 minutes after drug intake | 1.7 (0.4) | 1.5 (0.5)
  3 hours after drug intake: number analyzed (Observations) | 91 | 45
  3 hours after drug intake | 1.4 (0.4) | 1.9 (0.6)
  4 hours after drug intake: number analyzed (Observations) | 91 | 45
  4 hours after drug intake | 2.5 (0.4) | 2.4 (0.5)
  8 hours after drug intake: number analyzed (Observations) | 91 | 45
  8 hours after drug intake | 6.0 (0.5) | 6.5 (0.7)
  12 hours after drug intake: number analyzed (Observations) | 91 | 45
  12 hours after drug intake | 11.6 (0.5) | 11.0 (0.7)
  24 hours after drug intake: number analyzed (Observations) | 91 | 45
  24 hours after drug intake | 6.9 (0.5) | 5.7 (0.6)
Statistical Analysis 1: Comparison: Placebo to BI 409306 in 2 Periods vs 50 Milligram (mg) BI 409306; [analysis description as in outcome 1, analysis 1]; Test type: Other — No formal hypotheses were tested; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Difference of adjusted means = 2.4, 90% CI 2-sided [1.4 to 3.3], Standard Error of Mean 0.6 — Maximum difference of adjusted means was calculated as BI 409306 - placebo at 20 minutes after drug intake

8. Secondary Outcome: Change From Baseline in Heart Rate (HR) at That Timepoint Between 20 Minutes to 24 Hours After Drug Administration Where the Difference of Means in Heart Rate Changes From Baseline Between 250 Milligram (mg) BI 409306 and Placebo Takes Its Maximum
Description: Change from baseline in heart rate (HR) at that timepoint between 20 minutes to 24 hours after drug administration where the difference of means in heart rate changes from baseline between 250 milligram (mg) BI 409306 and placebo takes its maximum.
  A linear mixed-effects model for repeated measurements based on Schall and Ring (MMRM) was fitted to the observations for 250 mg BI 409306 and the 2 placebo periods.
  Total number of participants per treatment and timepoint can be lower than 47 due to participants having left their treatment sequence before being exposed to the respective treatment, or due to exclusion of individual participant ECG data at timepoints affected by ECG-relevant important protocol deviations.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: beats / minute
Units Other Than Participants: Observations
Arm/Group | Placebo to BI 409306 in 2 Periods | 250 Milligram (mg) BI 409306
Number analyzed (Participants) | 47 | 46
Number analyzed (Observations) | 1000 | 505
beats / minute
  20 minutes (min) after drug intake: number analyzed (Participants) | 47 | 45
  20 minutes (min) after drug intake: number analyzed (Observations) | 90 | 45
  20 minutes (min) after drug intake | 0.6 (0.6) | 8.9 (0.8)
  40 min after drug intake = timepoint of maximum: number analyzed (Observations) | 91 | 46
  40 min after drug intake = timepoint of maximum | 0.3 (0.5) | 12.0 (0.6)
  1 hour after drug intake: number analyzed (Observations) | 91 | 46
  1 hour after drug intake | 0.4 (0.5) | 8.1 (0.6)
  1 hour and 30 minutes after drug intake: number analyzed (Observations) | 91 | 46
  1 hour and 30 minutes after drug intake | 0.6 (0.5) | 4.4 (0.6)
  2 hours after drug intake: number analyzed (Observations) | 91 | 46
  2 hours after drug intake | 0.8 (0.5) | 3.2 (0.6)
  2 hours and 30 minutes after drug intake: number analyzed (Observations) | 91 | 46
  2 hours and 30 minutes after drug intake | 1.6 (0.5) | 2.9 (0.6)
  3 hours after drug intake: number analyzed (Observations) | 91 | 46
  3 hours after drug intake | 1.4 (0.5) | 1.9 (0.6)
  4 hours after drug intake: number analyzed (Observations) | 91 | 46
  4 hours after drug intake | 2.4 (0.5) | 3.2 (0.6)
  8 hours after drug intake: number analyzed (Observations) | 91 | 46
  8 hours after drug intake | 5.9 (0.5) | 6.5 (0.7)
  12 hours after drug intake: number analyzed (Observations) | 91 | 46
  12 hours after drug intake | 11.5 (0.5) | 11.5 (0.7)
  24 hours after drug intake: number analyzed (Observations) | 91 | 46
  24 hours after drug intake | 6.8 (0.5) | 6.8 (0.6)
Statistical Analysis 1: Comparison: Placebo to BI 409306 in 2 Periods vs 250 Milligram (mg) BI 409306; [analysis description as in outcome 2, analysis 1]; Test type: Other — No formal hypotheses were tested; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Difference of adjusted means = 11.7, 90% CI 2-sided [10.6 to 12.8], Standard Error of Mean 0.7 — Maximum difference of adjusted means was calculated as BI 409306 - placebo at 40 minutes after drug intake

9. Secondary Outcome: Change From Baseline in Heart Rate (HR) at That Timepoint Between 20 Minutes to 24 Hours After Drug Administration Where the Difference of Means in Heart Rate Changes From Baseline Between 50 Milligram (mg) BI 409306 and Placebo Takes Its Minimum
Description: Change from baseline in heart rate (HR) at that timepoint between 20 minutes to 24 hours after drug administration where the difference of means in heart rate changes from baseline between 50 milligram (mg) BI 409306 and placebo takes its minimum.
  A linear mixed-effects model for repeated measurements based on Schall and Ring (MMRM) was fitted to the observations for 50 mg BI 409306 and the 2 placebo periods.
  Total number of participants per treatment and timepoint can be lower than 47 due to participants having left their treatment sequence before being exposed to the respective treatment, or due to exclusion of individual participant ECG data at timepoints affected by ECG-relevant important protocol deviations.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: beats / minute
Units Other Than Participants: Observations
Arm/Group | Placebo to BI 409306 in 2 Periods | 50 Milligram (mg) BI 409306
Number analyzed (Participants) | 47 | 45
Number analyzed (Observations) | 1000 | 493
beats / minute
  20 min after drug intake: number analyzed (Observations) | 90 | 45
  20 min after drug intake | 0.6 (0.4) | 3.0 (0.5)
  40 minutes after drug intake: number analyzed (Observations) | 91 | 45
  40 minutes after drug intake | 0.4 (0.4) | 2.5 (0.5)
  1 hour after drug intake: number analyzed (Observations) | 91 | 45
  1 hour after drug intake | 0.5 (0.4) | 1.9 (0.5)
  1 hour and 30 minutes after drug intake: number analyzed (Participants) | 47 | 43
  1 hour and 30 minutes after drug intake: number analyzed (Observations) | 91 | 43
  1 hour and 30 minutes after drug intake | 0.7 (0.4) | 0.8 (0.5)
  2 hours after drug intake: number analyzed (Observations) | 91 | 45
  2 hours after drug intake | 0.9 (0.4) | 0.8 (0.5)
  2 hours and 30 minutes after drug intake: number analyzed (Observations) | 91 | 45
  2 hours and 30 minutes after drug intake | 1.7 (0.4) | 1.5 (0.5)
  3 hours after drug intake: number analyzed (Observations) | 91 | 45
  3 hours after drug intake | 1.4 (0.4) | 1.9 (0.6)
  4 hours after drug intake: number analyzed (Observations) | 91 | 45
  4 hours after drug intake | 2.5 (0.4) | 2.4 (0.5)
  8 hours after drug intake: number analyzed (Observations) | 91 | 45
  8 hours after drug intake | 6.0 (0.5) | 6.5 (0.7)
  12 hours after drug intake: number analyzed (Observations) | 91 | 45
  12 hours after drug intake | 11.6 (0.5) | 11.0 (0.7)
  24 hours after drug intake = timepoint of minimum: number analyzed (Observations) | 91 | 45
  24 hours after drug intake = timepoint of minimum | 6.9 (0.5) | 5.7 (0.6)
Statistical Analysis 1: Comparison: Placebo to BI 409306 in 2 Periods vs 50 Milligram (mg) BI 409306; [analysis description as in outcome 1, analysis 1]; Test type: Other — No formal hypotheses were tested; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Difference of adjusted means = -1.2, 90% CI 2-sided [-2.3 to -0.1], Standard Error of Mean 0.6 — Minimum difference of adjusted means was calculated as BI 409306 - placebo at 24 hours after drug intake

10. Secondary Outcome: Change From Baseline in Heart Rate (HR) at That Timepoint Between 20 Minutes to 24 Hours After Drug Administration Where the Difference of Means in Heart Rate Changes From Baseline Between 250 Milligram (mg) BI 409306 and Placebo Takes Its Minimum
Description: Change from baseline in heart rate (HR) at that timepoint between 20 minutes to 24 hours after drug administration where the difference of means in heart rate changes from baseline between 250 milligram (mg) BI 409306 and placebo takes its minimum.
  A linear mixed-effects model for repeated measurements based on Schall and Ring (MMRM) was fitted to the observations for 250 mg BI 409306 and the 2 placebo periods.
  Total number of participants per treatment and timepoint can be lower than 47 due to participants having left their treatment sequence before being exposed to the respective treatment, or due to exclusion of individual participant ECG data at timepoints affected by ECG-relevant important protocol deviations.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: beats / minute
Units Other Than Participants: Observations
Arm/Group | Placebo to BI 409306 in 2 Periods | 250 Milligram (mg) BI 409306
Number analyzed (Participants) | 47 | 46
Number analyzed (Observations) | 1000 | 505
beats / minute
  20 min after drug intake: number analyzed (Participants) | 47 | 45
  20 min after drug intake: number analyzed (Observations) | 90 | 45
  20 min after drug intake | 0.6 (0.6) | 8.9 (0.8)
  40 minutes after drug intake: number analyzed (Observations) | 91 | 46
  40 minutes after drug intake | 0.3 (0.5) | 12.0 (0.6)
  1 hour after drug intake: number analyzed (Observations) | 91 | 46
  1 hour after drug intake | 0.4 (0.5) | 8.1 (0.6)
  1 hour and 30 minutes after drug intake: number analyzed (Observations) | 91 | 46
  1 hour and 30 minutes after drug intake | 0.6 (0.5) | 4.4 (0.6)
  2 hours after drug intake: number analyzed (Observations) | 91 | 46
  2 hours after drug intake | 0.8 (0.5) | 3.2 (0.6)
  2 hours and 30 minutes after drug intake: number analyzed (Observations) | 91 | 46
  2 hours and 30 minutes after drug intake | 1.6 (0.5) | 2.9 (0.6)
  3 hours after drug intake: number analyzed (Observations) | 91 | 46
  3 hours after drug intake | 1.4 (0.5) | 1.9 (0.6)
  4 hours after drug intake: number analyzed (Observations) | 91 | 46
  4 hours after drug intake | 2.4 (0.5) | 3.2 (0.6)
  8 hours after drug intake: number analyzed (Observations) | 91 | 46
  8 hours after drug intake | 5.9 (0.5) | 6.5 (0.7)
  12 hours after drug intake=timepoint of minimum: number analyzed (Observations) | 91 | 46
  12 hours after drug intake=timepoint of minimum | 11.5 (0.5) | 11.5 (0.7)
  24 hours after drug intake: number analyzed (Observations) | 91 | 46
  24 hours after drug intake | 6.8 (0.5) | 6.8 (0.6)
Statistical Analysis 1: Comparison: Placebo to BI 409306 in 2 Periods vs 250 Milligram (mg) BI 409306; [analysis description as in outcome 2, analysis 1]; Test type: Other — No formal hypotheses were tested; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Difference of adjusted means = -0.0, 90% CI 2-sided [-1.3 to 1.3], Standard Error of Mean 0.8 — Minimum difference of adjusted means was calculated as BI 409306 - placebo at 12 hours after drug intake

ADVERSE EVENTS:
Time Frame: On-treatment period, that is, from administration of study drug until the end of the respective Residual Effect Period (24 hours for BI 409306 and placebo, 4 days for moxifloxacin), up to 4 days.
Description: Treated set (TS): This participant set included all randomized participants who received at least one dose of any trial medication.
  Each treatment represents one period out of five treatment periods in the treatment sequences and only includes the total number of participants exposed to that treatment. Total number of participants per treatment is lower than number of participants in TS due to participants having left the sequence before being exposed to the respective treatment.
Groups:
- Placebo 1 to BI 409306: Placebo 1 to BI 409306 administered orally as a single dose (5 film-coated tablets) taken with 240 milliliter of water after an overnight fast of at least 10 hours on day 1 of the treatment period.
- Placebo 2 to BI 409306: Placebo 2 to BI 409306 administered orally as a single dose (5 film-coated tablets) taken with 240 milliliter of water after an overnight fast of at least 10 hours on day 1 of the treatment period.
Arm/Group | Placebo 1 to BI 409306 | Placebo 2 to BI 409306 | 50 Milligram (mg) BI 409306 | 250 Milligram (mg) BI 409306 | 400 Milligram (mg) Moxifloxacin
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/46 | 0/45 | 0/46 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/46 | 0/45 | 0/46 | 0/45
Other Adverse Events (participants affected / at risk) | 2/45 | 3/46 | 12/45 | 36/46 | 3/45
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo 1 to BI 409306 (N=45) | Placebo 2 to BI 409306 (N=46) | 50 Milligram (mg) BI 409306 (N=45) | 250 Milligram (mg) BI 409306 (N=46) | 400 Milligram (mg) Moxifloxacin (N=45)
Chromatopsia (Eye disorders) | 0 | 1 | 3 | 19 | 0
Photophobia (Eye disorders) | 0 | 1 | 4 | 14 | 0
Photopsia (Eye disorders) | 0 | 0 | 0 | 7 | 0
Visual brightness (Eye disorders) | 0 | 0 | 1 | 3 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 3 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 8 | 2
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 5 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 3 | 2 | 0
Headache (Nervous system disorders) | 1 | 1 | 3 | 7 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-04-23): https://cdn.clinicaltrials.gov/large-docs/03/NCT03934203/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-18): https://cdn.clinicaltrials.gov/large-docs/03/NCT03934203/SAP_001.pdf